CLINICAL TRIAL: NCT06383689
Title: Placebo Optimization of the Presurgical Long-term Video-EEG Monitoring (OPERA)
Brief Title: Placebo Optimization of the Presurgical Long-term Video-EEG Monitoring
Acronym: OPERA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Christian Hoppe, Senior Researcher (Clinical Neuropsychologist), University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Az. 297/23-EP
Record Dates: First submitted 2024-04-10; First posted 2024-04-25 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Symptomatic Epilepsy
Keywords: epilepsy; emotional well-being; placebo; video-EEG long-term monitoring; presurgical epilepsy diagnostics
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: monocentric single-blinded randomized clinical study on the effectiveness of covered placebo on epileptic seizure occurrence and emotional well-being with 3 study conditions: "seizure pill" (PCB-S), "well-being pill" (PCB-W) and no pill (control)
Who Masked: Participant
Masking Description: Like in psychological studies, only patients can participate in the study who consent to accept that complete study information can only be provided after the entire study was finished (with an option to withdraw consent at that point) as information on ingredients of the study pill (which is placebo) must be concealed for inherent reasons (study on effects of covered placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Seizure placebo pill (PCB-S) (Experimental): Patients assigned to this condition receive a covered placebo pill (1-0-1) on a daily basis with the indication of possible acceleration of the occurrence of an epileptic seizure (which then allows to conclude V-EEG monitoring faster)
  Interventions: Other: Seizure placebo pill
- Well-being placebo pill (PCB-W) (Experimental): Patients assigned to this condition receive a covered placebo pill (1-0-1) on a daily basis with the indication of possible improvement of emotional well-being during the demanding V-EEG monitoring procedure
  Interventions: Other: Well-being placebo pill
- No pill (control) (No Intervention): Patients assigned to this condition receive no study pill but are asked to fill-in all questionnaires and diaries like patients in the two active arms

INTERVENTIONS:
Other: Seizure placebo pill — patients in this study arm receive a covered placebo pill on a daily basis (1-0-1) with the indication of possible acceleration of seizure occurrence during presurgical video-EEG
  Other Names: PCB-S
  Arms: Seizure placebo pill (PCB-S)
Other: Well-being placebo pill — patients in this study arm receive a covered placebo pill on a daily basis (1-0-1) with the indication of possible improvement of emotional well-being during video-EEG
  Other Names: PCB-W
  Arms: Well-being placebo pill (PCB-W)

SUMMARY:
The notion of genuine placebo effects on epileptic seizure events (i.e., effects beyond methodological study artifacts) is incompatible with the standard model of epilepsy seizure genesis. In this single-blind controlled study, the effectiveness of a covered placebo on (1) the timing of the occurrence of a first epileptic seizure ("seizure pill") versus (2) the subjective well-being ("comfort pill") during pre-surgical video-EEG monitoring will be examined. It is hypothesized that a placebo effect on subjective well-being can be demonstrated, but that epileptic seizure events are not influenced by placebo.

DETAILED DESCRIPTION:
Patients undergoing long-term video-EEG monitoring for the purpose of pre-operative epilepsy diagnostics will be invited to participate in the study. Patients will be pseudo-randomized into three study conditions (in blocks of six). The study participants will take a placebo pill designated either as a "seizure pill" (Condition PCB-S) or a "comfort pill" (PCB-W) in addition to their regular medication in the morning and evening, or not receive any additional placebo medication (No-PCB).

Both the "seizure pill" and the "comfort pill" are commercially available, ingredient-free placebo pills (P-pills blue Lichtenstein, produced by Winthrop Pharmaceuticals). No further details about the composition of the pill will be provided; information about the ingredients of the respective pill will be provided after the end of the entire study. Depending on randomization, study participants will be informed that this pill is expected to (1) either facilitate/accelerate the occurrence of epileptic seizures (PCB-S) (thereby shortening the required time for video-EEG monitoring), or (2) to lead to a more stable/improved emotional well-being during the stay in the V-EEG (PCB-W) or (3) will not receive a pill but are asked to fill-in questionnaires and diaries like the other patients.Start of the V-EEG will be documented as the starting point for latency measurement for the occurrence of a first epileptic seizure. The patients will be pseudo-randomized into the three study conditions: Out of every 6 patients, 2 will be assigned to each of the three study conditions. Patients in both active study conditions will receive the first pill at the start of the V-EEG. After that, study participants will receive the respective "pill" morning and evening in addition to their other medications, however, visibly separated from them and clearly marked as study medication. All participants, including controls, will keep a seizure diary during the V-EEG. In addition, they will fill-in a newly constructed ad-hoc questionnaire at the beginning and after the V-EEG. Finally, all patients will be asked twice daily (around 9 AM and around 6 PM) about their overall emotional well-being using a visual analogue scale (VAS; 0 very bad ... 100 extremely good). The highly standardized clinical procedures of presurgical evaluation are in no way affected by the study. In particular, anti-seizure medications for all patients will be tapered off following exactly the same schedule without any influence from the study; the medication will be precisely documented.

ELIGIBILITY:
Inclusion Criteria:

* eligibility for presurgical epilepsy diagnostics

Exclusion Criteria:

* inclusion criterion implies all exclusion criteria for this procedure
* legal guardian
* lack of consent or lack of capability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Latency to first epileptic seizure | immediately after video-EEG monitoring
  temporal latency from beginning of the video-EEG monitoring to the occurrence of the first epileptic seizure

SECONDARY OUTCOMES:
Occurrence of an epileptic seizure | immediately after video-EEG monitoring
  Occurrence of an epileptic seizure during the video-EEG (yes/no)
Early occurrence of an epileptic seizure within the first 72 hours | immediately after video-EEG monitoring
  Early occurrence of an epileptic seizure within the first 72 hours of video-EEG monitoring (yes/no)
Number of epileptic seizures during the video-EEG | immediately after video-EEG monitoring
  Total number of epileptic seizures which occurred during the video-EEG
Number of early occurring epileptic seizures | 72 hours after video-EEG monitoring
  Total number of epileptic seizures recorded during the first 72 hours of video-EEG
Daily average frequency of epileptic seizures | immediately after video-EEG monitoring
  Average daily frequency of epileptic seizures during the entire video-EEG (calculated)
Very early first epileptic seizure | after 1st day after video-EEG monitoring
  First epileptic seizure on the first day of video-EEG (yes/no)
Early epileptic seizure | after 2nd day after video-EEG monitoring
  First epileptic seizure on the first or second day of video-EEG (yes/no)
Epileptic seizure within the first three days | after 3rd day after video-EEG monitoring
  First epileptic seizure within the first three days of video-EEG (yes/no).
Emotional well-being | immediately after video-EEG monitoring
  Visual analogue scales (diary), 2x daily queries (9 am, 6 pm): mean and standard deviation (stability), during the video-EEG
Dissociative non-epileptic seizures | immediately after video-EEG monitoring
  occurrence of dissociative non-epileptic seizures during video-EEG (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Surges, Prof., Principal Investigator — Department of Epileptology, University Hospital Bonn, Germany
Locations (1):
- Department of Epileptology, University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No